CLINICAL TRIAL: NCT02529007
Title: Endo-cuff Assisted Colonoscopy Versus Standard Colonoscopy for Polyp Detection in Bowel Cancer Screening Patients: A Randomised Controlled Trial. The E-CAP Study
Brief Title: Endo-cuff Assisted Vs. Standard Colonoscopy for Polyp Detection in Bowel Cancer Screening
Acronym: E-CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PHT/2013/71
Record Dates: First submitted 2015-07-17; First posted 2015-08-19 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2015-07

CONDITIONS: Colonic Polyps; Colonic Neoplasms
Keywords: Colonoscopy; early cancer detection; cancer screening
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (Active Comparator): These patients have standard colonoscopy performed
  Interventions: Other: Standard colonoscopy
- Endocuff (Experimental): These patients have colonoscopy performed with the endo-cuff attached to the end of the colonoscope
  Interventions: Device: Endo-cuff

INTERVENTIONS:
Device: Endo-cuff — Colonoscopy performed with endo-cuff attached to the colonoscope
  Arms: Endocuff
Other: Standard colonoscopy — Standard colonoscopy without end-cuff
  Arms: Standard

SUMMARY:
The study evaluates whether the use of a novel endoscopic cap (the endo-cuff) at the tip of a colonoscope improves the numbers of polyps detected during bowel cancer screening colonoscopy. Half the patients will have standard colonoscopy and half will have colonoscopy with the cap attached.

DETAILED DESCRIPTION:
Problem statement:

In England, everyone in the age group of 60-69 years is invited to participate in bowel cancer screening. Those who test positive in the initial screening stool test are invited to have a colonoscopy. The purpose of colonoscopy is to detect any obvious cancers, and in the absence of obvious cancers the purpose is to detect and remove all the polyps present in the colon, as polyps have the potential to develop into cancers. However, colonoscopy still misses up to 25% of polyps. Cap assisted colonoscopy improves polyp detection but still misses a significant number of polyps. There is a need for an improved cap design which will help improve polyp detection.

Research question/hypothesis:

Does using an endocuff on a colonoscope improve polyp detection as compared to standard colonoscopy in bowel cancer screening patients?

Study design:

Parallel group, single blinded randomised controlled trial

Study participants:

Patients attending for colonoscopy under the bowel cancer screening programme

Planned sample size: 534

Planned study period: 12 months

Primary objective:

To assess the impact of endocuff assisted colonoscopy on the number of polyps detected per patient

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for colonoscopy under the national bowel cancer screening programme
* Able to provide written informed consent

Exclusion Criteria:

* History of Inflammatory bowel disease
* History of Hereditary non polyposis colorectal cancer

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of polyps detected per patient | 1 month (when pathology report available)

SECONDARY OUTCOMES:
Cancer detection rate | 1 month (when pathology report available)
Polyp detection rate | 1 month (when pathology report available)
Adenomas per patient | 1 month (when pathology report available)
Adenoma detection rate | 1 month (when pathology report available)
Caecal intubation rate | 1 day
  will be recorded at the time of the procedure
Total procedure time - from scope insertion to removal | 1 day
  will be recorded at the time of the procedure
Time taken to reach caecum | 1 day
  will be recorded at the time of the procedure
Time taken to withdraw scope (from caecum to removal of scope) | 1 day
  will be recorded at the time of the procedure
Patient comfort score | 1 day
  will be recorded at the time of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MBBS, MD, MRCP, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Derived] Bhattacharyya R, Chedgy F, Kandiah K, Fogg C, Higgins B, Haysom-Newport B, Gadeke L, Thursby-Pelham F, Ellis R, Goggin P, Longcroft-Wheaton G, Bhandari P. Endocuff-assisted vs. standard colonoscopy in the fecal occult blood test-based UK Bowel Cancer Screening Programme (E-cap study): a randomized trial. Endoscopy. 2017 Nov;49(11):1043-1050. doi: 10.1055/s-0043-111718. Epub 2017 Jun 14. PMID 28614895